CLINICAL TRIAL: NCT02320708
Title: A Randomized, Double-Blind, Placebo- and Active- Controlled, Single-Dose, Efficacy, Safety, and Pharmacokinetics Proof of Concept Study of a Test Acetaminophen 500 mg Tablet in Postoperative Dental Pain
Brief Title: Study of Acetaminophen (ACE) in Post-operative Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc. (Industry)
Collaborators: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO-140128120904-PACT
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Dental Pain
Keywords: Molar,third; Teeth,wisdom; Pain, Postoperative; Dental Surgery; Third molar extraction
MeSH Terms: conditions — Toothache; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test Acetaminophen (ACE) (1000 mg) and placebo (Experimental)
  Interventions: Drug: Acetaminophen (ACE) (1000 mg); Drug: Placebo
- Commerical ACE (1000 mg) and placebo (Active Comparator)
  Interventions: Drug: Commercial ACE (1000 mg); Drug: Placebo
- Commerical Ibuprofen (IBU) (400 mg) and placebo (Active Comparator)
  Interventions: Drug: Commercial Ibuprofen (IBU) (400 mg); Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen (ACE) (1000 mg) — 2 Test ACE 500 mg tablets taken orally one time
  Arms: Test Acetaminophen (ACE) (1000 mg) and placebo
Drug: Commercial ACE (1000 mg) — 2 ACE 500 mg caplets taken orally one time
  Arms: Commerical ACE (1000 mg) and placebo
Drug: Commercial Ibuprofen (IBU) (400 mg) — 2 IBU 200 mg soft-gels taken orally one time
  Arms: Commerical Ibuprofen (IBU) (400 mg) and placebo
Drug: Placebo — 2 placebo caplets for acetaminophen taken orally one time
  Arms: Commerical Ibuprofen (IBU) (400 mg) and placebo; Placebo; Test Acetaminophen (ACE) (1000 mg) and placebo
Drug: Placebo — 2 placebo soft-gels for ibuprofen taken orally one time
  Arms: Commerical ACE (1000 mg) and placebo; Placebo; Test Acetaminophen (ACE) (1000 mg) and placebo
Drug: Placebo — 2 placebo tablets for Test acetaminophen taken orally one time
  Arms: Commerical ACE (1000 mg) and placebo; Commerical Ibuprofen (IBU) (400 mg) and placebo; Placebo

SUMMARY:
This is a dental pain study evaluating the efficacy and safety of a single dose of test acetaminophen (ACE) (1000 mg) compared to commercial acetaminophen (1000 mg), ibuprofen (IBU) (400 mg), and placebo over a 6 hour period. Subjects will undergo dental extraction of three or four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. Are 17 to 50 years of age
2. Weigh 100 lbs or greater and body mass index (BMI) 18 to 30 (inclusive)
3. Dental extraction of three or four third-molars.
4. Experience moderate to severe pain after extraction of third molars

Exclusion Criteria:

1. Currently pregnant (or planning to be pregnant) or nursing a baby
2. Known allergy to acetaminophen (ACE) or non-steroidal anti-inflammatory drugs (NSAIDs)
3. Inability to swallow whole large tablets or capsules
4. Have other conditions that the investigator feels may impact subject's safety and/or the integrity of the study

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Time weighted sum of pain intensity difference from 0-6 hours (SPID 0-6) | 6 Hours
  Time weighted sum of pain intensity difference scores from baseline over 6 hours. Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain

SECONDARY OUTCOMES:
Time weighted sum of pain intensity difference from 0-4 hours (SPID 0-4) | 4 Hours
  Time weighted sum of pain intensity difference scores from baseline over 4 hours. Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Time to meaningful pain relief | Within 6 Hours
  Minutes until meaningful pain relief are achieved. Stopwatch is started after the subject takes the study medication. The subjects are instructed to stop the stopwatch when the relief from the starting pain is meaningful to them.
Time to first perceptible pain relief | Within 6 Hours
  Minutes until first perceptible pain relief is achieved. Stopwatch is started after the subject takes the study medication. The subject is instructed to stop the stopwatch when they first begin to feel any pain relief.
Time to confirmed first perceptible relief | Within 6 Hours
  Minutes until confirmed first perceptible pain relief are achieved. Stopwatch is started after the subject takes the study medication. The subject is instructed to stop the stopwatch when they first begin to feel any pain relief. The first perceptible pain relief is confirmed if the subject also stopped the second stopwatch indicating meaningful pain relief.
Time weighted sum of pain relief from 0-4 (TOTPAR 0-4) | 4 hours
  Time weighted sum of pain relief scores over four hours. Pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Time weighted sum of pain relief from 0-6 (TOTPAR 0-6) | 6 hours
  Time weighted sum of pain relief scores over six hours. Pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Duration of relief after dosing (time to rescue analgesic) | 6 Hours
  Minutes until rescue medication is given
Proportion of subjects taking a rescue analgesic by 6 hours | 6 Hours
  Percentage of subjects using rescue medication through six hours
Subject Global Evaluation assessed at hour 6 or at time of rescue | 6 hours
  Patient assessment of the pain medication - number of subjects rating the medication they received as a pain reliever on a score of 0-4, where 0=poor, 1=fair, 2=good, 3=very good, 4=excellent
Pain relief (PAR) scores at 0.25 Hours | 0.25 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 0.5 Hours | 0.5 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 0.75 Hours | 0.75 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 1 Hours | 1 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 1.25 Hours | 1.25 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 1.5 Hours | 1.5 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 2 Hours | 2 hoursH
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 3 Hours | 3 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 4 Hours | 4 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 5 Hours | 5 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain relief (PAR) scores at 6 Hours | 6 Hours
  Pain relief scores at each assessment time point - pain relief was evaluated using a 0-10 pain relief numerical rating scale (PR-NRS) where 0 = no relief and 10 = complete relief
Pain intensity difference (PID) at 0.25 Hours | 0.25 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 0.5 Hours | 0.5 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 0.75 Hours | 0.75 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 1 Hours | 1 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 1.25 Hours | 1.25 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 1.5 Hours | 1.5 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 2 Hours | 2 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 3 Hours | 3 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 4 Hours | 4 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 5 Hours | 5 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain
Pain intensity difference (PID) at 6 Hours | 6 Hours
  Pain intensity difference (PID) from baseline at each assessment time point - Pain intensity was evaluated using a 0-10 pain intensity numerical rating scale (PI-NRS) where 0 = no pain and 10 = very severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided